CLINICAL TRIAL: NCT00793507
Title: Oral Health Care Early Intervention Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Delta Dental Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-0198; PN200703-001 (Other Grant/Funding Number: Delta Dental)
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2009-01

CONDITIONS: Caries
Keywords: childhood caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Intervention Group (Experimental): All participants in the intervention group will be receiving standard preventive dental care received by children in their dental providers' office. These intervention children will receive dental scaling, cleaning and fluoride varnish at visits every three to six months. All participants in the intervention group will receive active reminder/recall from the hygienist, encouraging the participants to return every three to six months for the oral exam, cleaning, scaling and fluoride application.
  Interventions: Other: Oral Health Care Early Intervention Project
- 2: Control Group (Active Comparator): The control group will receive usual care, but will not receive pre-scheduling, reminders, or care coordination by the dental hygienist.
  Interventions: Other: Oral Health Care Early Intervention Project

INTERVENTIONS:
Other: Oral Health Care Early Intervention Project — The intervention group will receive routine preventive dental care, 2 to 4 times per year depending on risk of caries. The intervention group will also receive pre-scheduling, reminders, and care coordination by the dental hygienist. The control group will receive usual care, but will not receive pre-scheduling, reminders, or care coordination by the dental hygienist. In order to determine the incidence of early childhood caries at study enrollment, both intervention and control groups will receive a standardized oral examination with an assessment of caries presence and extent on the day of enrollment, at 12 months and at 24 months after enrollment. Both children in the control group and intervention group will be referred to a dentist if found to need restorative care.

SUMMARY:
This pilot project consists of co-locating dental hygienist services in medical primary care offices. Dental hygienists will work in close collaboration with the primary care offices, providing preventive dental care to young children either before or after scheduled well-child visits.

DETAILED DESCRIPTION:
This investigation is designed to determine the effect of having co-located dental hygienists in primary care offices on the incidence of early childhood caries among young children seen at these primary care offices. The dental hygienists will provide routine preventive dental care and oral health education within the usual scope of their practice. The study is also designed to assess parent knowledge, attitudes, and beliefs about oral health and perceived barriers to preventive dental care, as well as how their oral health-related attitudes change over time.

The specific aims for this project are:

Specific Aim 1: Among parents of young children seen in pediatric and family medicine primary care practices, determine the knowledge, attitudes, and beliefs of parents regarding the importance of oral health, means of preventing caries, and perceived barriers to accessing regular preventive dental care.

Specific Aim 2: After co-locating dental hygienists within pediatric and family medicine primary care practices, determine by randomized controlled trial the effect of routine preventive dental care provided by dental hygienists on the incidence of early childhood caries.

Specific Aim 3: Among parents of young children seen in pediatric and family medicine primary care practices, determine how parental oral health-related knowledge, attitudes, beliefs, and perceived barriers change over time, among parents of children seen by a co-located dental hygienist.

The major hypotheses for this project are:

1. Parents of children with public health insurance (Medicaid or Child Health Plan-Plus) will have one-half the odds of reporting a usual source of preventive dental care compared to children with private health insurance.
2. Among young children receiving routine preventive dental care by a co-located dental hygienist, 10% will develop dental caries over a 24-month period, compared with 20% caries experience among children who do not receive routine preventive dental care by a co-located dental hygienist.
3. Parents of children with early childhood caries (any caries in a primary tooth) which developed over a 24-month period will have more than twice the odds of reporting barriers to accessing a dental provider than parents of children with no early childhood caries.

ELIGIBILITY:
Inclusion Criteria:

Children with the following characteristics will be included in the study:

1. 0 - 36 months;
2. Have at least one tooth;
3. Have had one or more visits to a study practice in the prior 18 months.

Exclusion Criteria:

Children with the following characteristics will be excluded from the study:

1. No teeth; in essence child has not had any teeth erupt yet;
2. Chronic medical condition affecting oral health or the ability to perform routine preventive dental care, such as cerebral palsy, mental retardation, ectodermal dysplasia, and other genetic syndromes affecting oral health
3. Reports receiving primary health care somewhere else other than at one of the study practices;
4. Parents < 18 years of age.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1178 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
New ECC*(presence/absence) | At end of study, 24 months

SECONDARY OUTCOMES:
Association of ECC with perceived barriers to accessing a dental provider. | Day 1 of entry into study
Changes in parental knowledge, attitude, beliefs and barriers from pre- to post-study | At end of study, 24 months
Frequencies of parental knowledge, attitudes, beliefs and barriers (Descriptive variables: scales constructed of 4-point Likert items | Day 1 of entry into study
Severity of caries( presence/absence of S-ECC) | At end of study, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew F. Daley, MD, Principal Investigator — University of Colorado, Denver; Patricia Braun, MD, Study Director — University of Colorado, Denver
Locations (5):
- United States (5):
  - Rocky Mountain Youth, Aurora, Colorado
  - Grand Mesa Dental Hygiene, LLC, Delta, Colorado
  - Salud Family Health Centers, Fort Collins, Colorado
  - The Pediatric Associates, Montrose, Colorado
  - Rocky Mountain Youth, Thornton, Colorado

REFERENCES:
- [Background] Beltran-Aguilar ED, Barker LK, Canto MT, Dye BA, Gooch BF, Griffin SO, Hyman J, Jaramillo F, Kingman A, Nowjack-Raymer R, Selwitz RH, Wu T; Centers for Disease Control and Prevention (CDC). Surveillance for dental caries, dental sealants, tooth retention, edentulism, and enamel fluorosis--United States, 1988-1994 and 1999-2002. MMWR Surveill Summ. 2005 Aug 26;54(3):1-43. PMID 16121123
- [Background] U.S. Department of Health and Human Services. Oral Health in America: A Report of the Surgeon General. 1-332. 2000. Rockville, MD, U.S. Department of Health and Human Services, National Institute of Dental and Craniofacial Research, National Institutes of Health. Ref Type: Report
- [Background] Yu SM, Bellamy HA, Kogan MD, Dunbar JL, Schwalberg RH, Schuster MA. Factors that influence receipt of recommended preventive pediatric health and dental care. Pediatrics. 2002 Dec;110(6):e73. doi: 10.1542/peds.110.6.e73. PMID 12456940
- [Background] Kenney GM, McFeeters JR, Yee JY. Preventive dental care and unmet dental needs among low-income children. Am J Public Health. 2005 Aug;95(8):1360-6. doi: 10.2105/AJPH.2004.056523. PMID 16043667
- [Background] Liu J, Probst JC, Martin AB, Wang JY, Salinas CF. Disparities in dental insurance coverage and dental care among US children: the National Survey of Children's Health. Pediatrics. 2007 Feb;119 Suppl 1:S12-21. doi: 10.1542/peds.2006-2089D. PMID 17272579
- [Background] Edelstein BL. Disparities in oral health and access to care: findings of national surveys. Ambul Pediatr. 2002 Mar-Apr;2(2 Suppl):141-7. doi: 10.1367/1539-4409(2002)0022.0.co;2. PMID 11950385
- [Background] Lewis CW, Johnston BD, Linsenmeyar KA, Williams A, Mouradian W. Preventive dental care for children in the United States: a national perspective. Pediatrics. 2007 Mar;119(3):e544-53. doi: 10.1542/peds.2006-1958. PMID 17332174
- [Background] dela Cruz GG, Rozier RG, Slade G. Dental screening and referral of young children by pediatric primary care providers. Pediatrics. 2004 Nov;114(5):e642-52. doi: 10.1542/peds.2004-1269. PMID 15520094
- [Background] Lewis CW, Grossman DC, Domoto PK, Deyo RA. The role of the pediatrician in the oral health of children: A national survey. Pediatrics. 2000 Dec;106(6):E84. doi: 10.1542/peds.106.6.e84. PMID 11099627
- [Background] Mofidi M, Rozier RG, King RS. Problems with access to dental care for Medicaid-insured children: what caregivers think. Am J Public Health. 2002 Jan;92(1):53-8. doi: 10.2105/ajph.92.1.53. PMID 11772761
- [Background] Siegal MD, Marx ML, Cole SL. Parent or caregiver, staff, and dentist perspectives on access to dental care issues for head start children in Ohio. Am J Public Health. 2005 Aug;95(8):1352-9. doi: 10.2105/AJPH.2004.054858. Epub 2005 Jul 7. PMID 16006416
- [Background] Kelly SE, Binkley CJ, Neace WP, Gale BS. Barriers to care-seeking for children's oral health among low-income caregivers. Am J Public Health. 2005 Aug;95(8):1345-51. doi: 10.2105/AJPH.2004.045286. PMID 16043666
- [Background] Finlayson TL, Siefert K, Ismail AI, Delva J, Sohn W. Reliability and validity of brief measures of oral health-related knowledge, fatalism, and self-efficacy in mothers of African American children. Pediatr Dent. 2005 Sep-Oct;27(5):422-8. PMID 16435644
- [Background] American Academy of Pediatric Dentistry; American Academy of Pediatrics; American Academy of Pediatric Dentistry Council on Clinical Affairs. Policy on early childhood caries (ECC): classifications, consequences, and preventive strategies. Pediatr Dent. 2005-2006;27(7 Suppl):31-3. No abstract available. PMID 16541878
- [Background] Truman BI, Gooch BF, Sulemana I, Gift HC, Horowitz AM, Evans CA, Griffin SO, Carande-Kulis VG; Task Force on Community Preventive Services. Reviews of evidence on interventions to prevent dental caries, oral and pharyngeal cancers, and sports-related craniofacial injuries. Am J Prev Med. 2002 Jul;23(1 Suppl):21-54. doi: 10.1016/s0749-3797(02)00449-x. PMID 12091093